CLINICAL TRIAL: NCT02965950
Title: Treatment of Patients With Advanced Breast Cancer Harboring TP53 Mutations With Dose-dense Cyclophosphamide - the p53 Breast Cancer Trial
Brief Title: The p53 Breast Cancer Trial
Acronym: p53b
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/816; 2016-003459-31 (EudraCT Number)
Record Dates: First submitted 2016-11-04; First posted 2016-11-17 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Breast Cancer; Metastatic Breast Carcinoma
Keywords: breast cancer; TP53; cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TP53 mutated, LABC (Experimental): Patients with locally advanced breast cancer, TP53 mutated disease. Dose-dense cyclophosphamide, after taxanes +/- anthracyclines.
  Interventions: Drug: Cyclophosphamide
- TP53 mutated, MBC, first line (Experimental): Patients with metastatic breast cancer, TP53 mutated disease. Dose-dense cyclophosphamide first line metastatic disease
  Interventions: Drug: Cyclophosphamide
- TP53 wt, LABC (Experimental): Patients with locally advanced breast cancer, TP53 wt disease. Dose-dense cyclophosphamide, after taxanes and anthracyclines.
  Interventions: Drug: Cyclophosphamide
- TP53 wt, MBC (Experimental): Patients with metastatic breast cancer, TP53 wt disease. Dose-dense cyclophosphamide, after taxanes and anthracyclines.
  Interventions: Drug: Cyclophosphamide
- TP53 mutated, MBC (Experimental): Patients with metastatic breast cancer, TP53 mutated disease. Dose-dense cyclophosphamide, after taxanes +/- anthracyclines.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — I.v. infusion
  Other Names: ATC-number: L01A A01

SUMMARY:
This is a multicenter, open labeled, phase 2 clinical trial, where patients are stratified to one of two treatment groups based on upfront TP53 mutation status; i.e. TP53 mutated vs. TP53 wt disease, and treated with dose-dense cyclphosphamide. Furthermore, patients included are stratified based on tumor stage; i.e. locally advanced breast cancer (M0 disease) or metastatic breast cancer (M1 disease). All participating cancer centers will prospectively include patients with breast cancer fulfilling the inclusion criteria.

If patients do not respond to the experimental treatment as outlined in the protocol, treatment with dose-dense cyclophosphamide will be terminated, and further cancer treatment will continue at the treating oncologist's discretion. The response data for all patients who have received at least one chemotherapy course will be included in the final efficacy analysis.

Tumor tissue, blood samples and radiology data will be collected before therapy starts, if therapy needs to be changed, and for patients with locally advanced breast cancer: at surgery. Response data will be evaluated closely during treatment, with clinical assessment of tumor size every two weeks for patients with locally advanced breast cancer and by radiology every eight weeks for patients with metastatic breast cancer. Evaluation of side effects/tolerance will be performed at every clinical visit, i.e. every two weeks for all patients included in the p53 trial.

DETAILED DESCRIPTION:
Stage IV breast cancer (distant metastases) remains a non-curable condition; thus, treatment is considered palliative. However, many patients may live for years with their metastatic disease with a reasonably good quality of life. As for locally advanced primary breast cancers in need of primary medical therapy, lack of responsiveness to regular chemotherapy is associated with a poor prognosis, with a high risk of relapse and, subsequent, breast cancer death. TP53 mutations have been shown to predict a poor response to anthracyclines, a group of cytotoxic agents which is extensively used and which is in general efficacious in breast cancer. Notably, dose-intensification with cyclophosphamide has been found to significantly improve the response rate in TP53 mutated primary breast cancers. Our preliminary experience indicates that the use of dose-dense cyclophosphamide monotherapy every 2nd week with G-CSF support is well tolerated. As for patients with metastatic disease for whom the alternative would be to receive continuous chemotherapy at 3-weekly intervals the hypothesis is that cyclophosphamide given at 2-weekly intervals over a limited time period, followed by a "treatment holiday" among responders should be associated with a non-inferior quality of life all-over. As for patients with TP53 mutated locally advanced breast cancers where standard chemotherapy fails, the hypothesis is that cyclophosphamide dose dense treatment may be an effective treatment option downstaging the tumor prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced breast cancers in need of pre-surgical chemotherapy or metastatic breast cancer in need of chemotherapy.
* Resistance to endocrine therapy:

Either i) estrogen and progesterone negative tumor, or ii) harboring an estrogen and / or progesterone positive tumor where regular endocrine therapies have failed or where the treating physician finds endocrine therapy not indicated.

- Prior cancer therapy:

Metastatic disease:

First line treatment (amendment 2018):

No prior chemotherapy*. Prior endocrine therapy +/- CDK4/6 inhibitor or mTOR inhibitors is allowed if hormone receptor positive, HER2 negative disease.

Late-stage disease (approved protocol):

i) Prior exposure to and resistance to a taxane regimen**. ii) Prior exposure to and resistance to an anthracycline regimen** -mandatory only for patients with TP53 wt tumors.

LABC:

i) Prior exposure to and lack of response to to a taxane regimen**. ii) Prior exposure to and lack of response to an anthracycline regimen** - mandatory only for patients with TP53 wt tumors.

* Only for patients with TP53 mutated disease. Previous adjuvant chemotherapy, including alkylating agents (cyclophosphamide a.o.) and/or platinum, is allowed if completed >12 months prior to inclusion in the trial.

** In metastatic breast cancer resistance to taxanes/anthracyclines is defined as progressive disease (PD). In LABC lack of response is defined as stable disease (SD) after 4 courses of chemotherapy or PD. Breast cancer relapsing within 12 months subsequent to adjuvant taxanes or anthracyclines is considered resistant and re-exposure is not required prior to inclusion in the trial. This relates also to patients who could not receive proper taxane or anthracycline therapy due to side effects or other medical reasons.

* The primary tumor or at least one metastatic lesion must be available for biopsy collection at protocol inclusion. Notably; for patients with primary metastatic breast cancer, TP53 status should be determined in a metastatic deposit; tissue from the primary tumor may not substitute (this relates both to patients with synchronous and metachronous metastatic disease).
* Patients must have clinically and/or radiographically documented measurable breast cancer according to RECIST.
* WHO performance status 0-1
* Known tumor ER, PGR and HER2 status in the current situation, i.e. archival and historic breast cancer tissue can not be used for patients with relapse of the disease. However, patients can be included regardless of hormone receptor and HER2 status; in case such information lacks at inclusion, it may be analysed on the biopsy retrospectively.
* Age >18 years
* Radiology studies (CT thorax/abdomen and bone scintigraphy/bone scan) and ecco cor must be performed within 28 days prior to start of treatment.
* Before patient registration, written informed consent must be given according to national and local regulations.
* Blood test requirements:
* Neutrophils > 1.0 x 109/L
* Platelets > 75 x 109/L
* Bilirubin < 20 µmol/L.
* Serum creatinine < 1.5 x ULN

Exclusion Criteria:

* Co-morbidity that, based on the assessment of the treating physician, may preclude the use of cyclophosphamide at actual doses.
* Psychological, familial, sociological or geographical condition(s) potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Pregnant or lactating patients.
* Clinical evidence of serious coagulopathy. Prior arterial/venous thrombosis or embolism does not exclude patients from inclusion, unless patient is considered unfit by study oncologist.
* Active cystitis (to be treated upfront)
* Active bacterial infections
* Urinary obstruction
* Known hypersensitivity towards cyclophosphamide or pegfilgrastim, their metabolites and other ingredients in the drug administration formulation.
* Patient not able to give an informed consent or comply with study regulations as deemed by study investigator.
* Amendment 2018: Patients with HER2 positive, metastatic breast cancer in the first line setting (Arm C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) measured clinically (with calipers) or radiologically per RECIST guidelines. | Four years
  ORR of dose dense cyclophosphamide in patients with TP53 mutated breast cancer or TP53 wt breast cancer.

SECONDARY OUTCOMES:
Number of patients harboring the same molecular aberration or set of aberrations, and which are associated with either response to treatment or survival. | Four years
  These are genomic and proteomic aberrations beyond TP53 mutations.
Number of patients harboring the same TP53 mutation subtype | Four years
  Assess whether responses are recorded among patients harbouring TP53 mutations belonging to particular mutation subgroups.
Number of patients achieving pathological complete response (pCR) | Four years
  Patients achieving pathological complete response (pCR), measured as no remaining infiltrative carcinoma in the breast and axillary nodes by histology, in TP53 wt and mutated subgroups, after dose-dense cyclophosphamide.
Recurrence-free survival | 14 years
  Recurrence-free survival after dose-dense cyclophosphamide.
Overall survival | 14 years
  Recurrence-free and overall survival after dose-dense cyclophosphamide.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Four years
  Safety and tolerability of dose-dense cyclophosphamide

CONTACTS AND LOCATIONS:
Overall Officials: Hans Petter Eikesdal, MD PhD, Principal Investigator — Haukeland University Hospital
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen, Hordaland
  - St. Olavs Hospital, Trondheim, Sør Trøndelag
  - Akershus University Hospital, Lørenskog
  - Stavanger University Hospital, Stavanger
  - University Hospital of Northern Norway, Tromsø

IPD SHARING:
Plan to Share IPD: Yes
Plan to share with collaborators